CLINICAL TRIAL: NCT05161520
Title: Impact of Capsular Tension Ring Implantation on Intraocular Lens Tilt and Decentration in Cataract Patients With High Myopia: a Randomized Controlled Trial
Brief Title: Impact of Capsular Tension Ring Implantation on Intraocular Lens Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuhua Tan (Other)
Responsible Party: Sponsor-Investigator, Xuhua Tan, Associate Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Organization: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021KYPJ128
Record Dates: First submitted 2021-12-02; First posted 2021-12-17 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Cataract; High Myopia
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IOL plus CTR Patients will undergo phacoemulsification combined with IOL and CTR implantation. (Active Comparator)
  Interventions: Procedure: phacoemulsification combined with IOL and CTR implantation
- single IOL Patients will undergo phacoemulsification combined with IOL implantation. (Placebo Comparator)
  Interventions: Procedure: phacoemulsification combined with IOL implantation

INTERVENTIONS:
Procedure: phacoemulsification combined with IOL and CTR implantation — Device: CTR (276001G； OPHTEC BV, Netherlands) Device: IOL (920H; Rayner Intracular Lenses Limited，Hove，East Sussex，UK) All patients undergo uneventful phacoemulsification by a 3.0 mm temporal transparent corneal incision using Centurion Vision System (Alcon Laboratories, Fort Worth, TX, USA). After the nucleus and cortex are removed, a capsular tension ring is implanted in the capsular bag and then IOL is implanted.
  Arms: IOL plus CTR Patients will undergo phacoemulsification combined with IOL and CTR implantation.
Procedure: phacoemulsification combined with IOL implantation — Device: IOL (920H; Rayner Intracular Lenses Limited，Hove，East Sussex，UK) All patients undergo uneventful phacoemulsification by a 3.0 mm temporal transparent corneal incision using Centurion Vision System (Alcon Laboratories, Fort Worth, TX, USA). After the nucleus and cortex are removed, IOL is implanted in the capsular bag.
  Arms: single IOL Patients will undergo phacoemulsification combined with IOL implantation.

SUMMARY:
This is a randomized controlled trial to investigate the effect of capsular tension ring (CTR) implantation on intraocular lens (IOL) tilt and decentration in cataract patients with high myopia.

DETAILED DESCRIPTION:
Exact positioning and alignment of the IOL with the visual axis are the prerequisites of high-quality visual performance after cataract surgery. A certain degree of IOL tilt and decentration occur after uneventful cataract surgery, most of which are clinically tolerant. However, the relatively large capsular bag volume, zonular weakness, and vitreous liquefaction in cataract patients with high myopia may increase the IOL position instability, such as tilt, decentration and even dislocation, leading to the deterioration of visual function. Thus, how to improve the long-term stability of IOL position in high myopic cataract patients is an urgent issue to be addressed.

Previous studies have shown that CTR implantation during cataract surgery can increase the IOL stability in patients with normal axial length; however, its impact on IOL position of cataract patients with high myopia remains unclear.

In this randomized clinical trial, patients who meet the inclusion criteria will be divided into three layers according to the axial length:

(1)26mm≤AL<28mm (2)28mm≤AL<30mm (3)AL≥30mm

We are going to recruit 186 patients in total, with 62 patients in each layer. Patients on each layer will be randomly divided into experimental group (CTR implantation) and control group (only IOL implantation). If both eyes of a patient meet the inclusion criteria, only the first operated eye is included in the statistics analysis.

All included patients will be followed up at 1 week, 1 month, 3 months, 6 months, and 1 year postoperatively. Visual acuity, IOL tilt, IOL decentration, posterior capsule attachment with IOL, anterior capsule contraction, posterior capsular opacification, and visual quality will be measured and compared between the experimental group and the control group at different timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old;
2. axis length≥26mm;
3. Visually significant cataract;
4. The patient is willing and able to complete all necessary follow-ups and examinations.

Exclusion Criteria:

1. Intraoperative or postoperative complications: such as intraoperative posterior capsular rupture, zonular dehiscence, secondary glaucoma, endophthalmitis, etc.;
2. Other ocular comorbidity: such as keratopathy, glaucoma, uveitis, retinopathy, lens dislocation and ocular trauma, etc.;
3. History of intraocular surgery;
4. Severe systemic diseases: such as severe hypertension, diabetes, heart disease, Alzheimer's, Parkinson, etc.;
5. Any condition that the study physician considers to be an impediment to the clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
IOL dencentration | 3 months after surgery
  Measured by anterior segment OCT (CASIA2)

SECONDARY OUTCOMES:
IOL dencentration | Baseline (before surgery), 1 week, 1 month, 6 months, 1 year after surgery
  Measured by anterior segment OCT (CASIA2)
IOL tilt | Baseline (before surgery), 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  Measured by anterior segment OCT (CASIA2)
Anterior capsule contraction | Baseline, 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  Compare the area of anterior capsule opening recorded by slit lamp photograph and analyzed by Image J software.
Posterior capsule attachment with IOL | 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  Measured by anterior segment OCT (CASIA2) and analyzed by Image J software.
Posterior capsular opacification | 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  Recorded by slit lamp photograph and analyzed by EPCO2000 analysis software.
BCVA | Baseline (before surgery), 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  BCVA is evaluated with ETDRS visual acuity chart.
Optical quality | Baseline (before surgery), 1 week, 1 month, 3 months, 6 months, 1 year after surgery
  Measured by OPD-SCAN III.
Visual function | 3 months, 6 months, 1 year after surgery
  Measured by visual function assessment questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin H, Zhang J, Jin A, Zhang Y, Zhang Y, Jin L, Xu Y, Xie X, Qiu X, Dai B, Tan X, Luo L, Liu Y. Capsular Tension Ring Implantation for Intraocular Lens Power Calculation in Highly Myopic Eyes: Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2025 May 1;143(5):373-381. doi: 10.1001/jamaophthalmol.2025.0110. PMID 40111331
- [Derived] Lin H, Zhang J, Zhang Y, Jin A, Zhang Y, Jin L, Xu Y, Xie X, Tan X, Luo L, Liu Y. Capsular Tension Ring Implantation for Intraocular Lens Decentration and Tilt in Highly Myopic Eyes: A Randomized Clinical Trial. JAMA Ophthalmol. 2024 Aug 1;142(8):708-715. doi: 10.1001/jamaophthalmol.2024.2215. PMID 38935400